CLINICAL TRIAL: NCT05519761
Title: A Retrospective, Observational, Multicenter Study to Evaluate the Safety and Performance of POLYSITE® and SEESITE® Implantable Ports
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Perouse Medical (Industry)
Collaborators: Eclevar Medtech (Industry)
Responsible Party: Sponsor
Other Study IDs: PSSS-2021-MULTI
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Veinous; Chemotherapy; Antibiotics; Antiviral Drugs; Parenteral Nutrition; Blood Transfusion; Blood Derivatives Transfusion; PMCF Study
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Implantation of veinous access ports — The surgeon, anaesthetist and interventional radiologist should be thoroughly familiar with the surgical procedure, instruments, and device characteristics prior to performing the implantation.
  The nurse has also to be familiar with the implantable port since he/she intervenes in it at the time of the Huber needle puncture and solution injection.

SUMMARY:
The purpose of this study is to evaluate performance and safety of POLYSITE® and SEESITE® implantable ports allowing repeated and prolonged access to the venous system for the administration of chemotherapy, antibiotics, antiviral drugs, parenteral nutrition, and for blood transfusion or blood derivatives transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Adult and paediatric population
* Patient who received the implantation of any POLYSITE® or SEESITE® implantable port referenced in the Annex 1 of the current protocol between 1-JAN-2018 and 31-DEC-2020

Exclusion Criteria:

* Patient who refused the data collection according to GDPR regulation applicable in France
* Patient who received the implantation of another device than those presented in Annex 1 of the current protocol.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All references of POLYSITE® and SEESITE® implantable ports apply to adult targeted population group.
  Only POLYSITE® and SEESITE® implantable ports referenced as 2000 series (micro size) and connected to a 5F catheter apply to paediatric (>10 kg) targeted population groups.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Performance : success of the insertion and placement of the implantable port. | Peri-procedure
  evaluation of the success of the insertion and placement of the implantable port.
Associate Performance : correct device insertion assess by Radiological endpoint | Peri-procedure
  percentage of patients with correct insertion into venous access objectively assessed via radiography, ECG or echography measurement
Associate Performance : correct device insertion assess Clinical endpoint | Peri-procedure
  percentage of patients with correct placement objectively assessed by clinical observation
Per-procedure Safety | 30 Days
  evaluation of the safety of the implantable ports
Associated Safety : rate of complications | 30 days
  measurement of the rate of complications reported during the short-term period of 30 days after the implantation date. As example, the following short-term complications will be looked at: infections, bleeding and hematoma, pneumothorax, hemothorax and pleural effusion, pain.

SECONDARY OUTCOMES:
Performance : evaluation of the device performance | 5 years
  percentage of patients with correct device insertion by the general surgeon, anaesthetist, or the radiologist. The insertion could be done under Echo or under fluoroscopy or ECG
device failure | 5 years
  measurement of the rate of device failure throughout the study until the device is removed from the patient's body. The device failures are defined as mechanical dysfunctions (catheter fracture, occlusion, and port-pocket dehiscence, pinch-off, embolization, leak, port/catheter disconnection, drug extravasation, mal-position, flip-over, migration, local venous thrombosis, etc…).
Safety: perioperative time | 5 years
  duration between the implantation procedure and the first use of the implantable port
Safety FU period: Device Failure Removal | 5 years
  the complications will be followed up to 30 days after the implantable port removal. If the removal is related to a device failure or a complication related to the device, the patient's safety will be followed until the resolution of the complication.the complications will be followed up to 30 days after the implantable port removal. If the removal is related to a device failure or a complication related to the device, the patient's safety will be followed until the resolution of the complication.
Safety Long Term period: Device Failure Removal | 5 years
  the complications will be followed up to 30 days after the implantable duration starting after the first 30 days after the implantation procedure and up to device removal, or patient death, or lost to follow-up, depending on what event comes first in the patient's medical chart. Study timepoints have been defined as 6-months Follow-up after the Implantation procedure, 12-months Follow-up after the Implantation procedure, 24-months Followup after the Implantation procedure and 36-months Follow-up after the Implantation procedure.
Safety Long Term period: complications | 5 years
  measurement of the rate of complications reported during the whole study and at the defined study timepoints. As example, the following long-term complications will be looked at: infections, inflammation, skin disorders, catheter-related venous thrombosis, pinch-off.
Emergent Risks | 5 years
  AEs collection

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHR d'Orléans, Orléans
  - Hopital Foch, Suresnes
  - IGR, Villejuif